CLINICAL TRIAL: NCT07146711
Title: A Prospective, Randomised, Open Label, Multiple Dose, Two-treatment, Two-period, Two-sequence, Crossover Bioequivalence Study of Tamsulosin Hydrochloride 0.4 mg, Prolonged-release Tablets (Synthon Hispania SL, Spain) Versus the Reference Drug Omnic Ocas®, Tamsulosin Hydrochloride 0.4 mg, Prolonged-release Film-coated Tablets (Astellas Pharma Europe B.V., the Netherlands), in Healthy Adult Male Subjects, at Steady State
Brief Title: A Comparative Bioavalability Study of Tamsulosin 0.4 mg Prolonged-release Tablets Versus the Reference Drug Omnic Ocas®, Tabsulosine 0.4 mg Tablets in Healthy Adult Male Subjects, at Steady State
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Berlin-Chemie AG Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BCAM/23/Tam-BE/001
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adult Males Volunteers
Keywords: Bioequivalence; Tamsulosin
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, multiple-dose, two-period, two-treatment, two-sequence crossover bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamsulosin hydrochloride 0.4 mg, prolonged-release tablets of Synthon Hispania SL, Spain (Experimental): Omnic Ocas®, Tamsulosin hydrochloride 0.4 mg, prolonged-release film-coated tablets of Astellas Pharma Europe B.V., the Netherlands
  Interventions: Drug: Tamsulosin (0.4 mg/j)
- Omnic Ocas®, Tamsulosin hydrochloride 0.4 mg, prolonged-release film-coated tablets of Astellas Phar (Active Comparator): Multiple dose administration (7 days)
  Interventions: Drug: Omnic Ocas®,

INTERVENTIONS:
Drug: Tamsulosin (0.4 mg/j) — Multiple dose administration (7 days)
  Arms: Tamsulosin hydrochloride 0.4 mg, prolonged-release tablets of Synthon Hispania SL, Spain
Drug: Omnic Ocas®, — Multiple dose administration (7 days)
  Arms: Omnic Ocas®, Tamsulosin hydrochloride 0.4 mg, prolonged-release film-coated tablets of Astellas Phar

SUMMARY:
The aim of this study is to evaluate the bioequivalence and safety of Tamsulosin hydrochloride 0.4 mg, prolonged-release tablets (Synthon Hispania SL, Spain), compared to Omnic Ocas®, Tamsulosin hydrochloride 0,4 mg, prolonged-release film-coated tablets (Astellas Pharma Europe B.V., the Netherlands), in healthy adult male subjects, at steady state.

DETAILED DESCRIPTION:
The assessment of the bioequivalence of Tamsulosin hydrochloride 0.4 mg, prolonged-release tablets (Synthon Hispania SL, Spain), and Omnic Ocas®, Tamsulosin hydrochloride 0.4 mg, prolonged-release film-coated tablets (Astellas Pharma Europe B.V., the Netherlands) after multiple dose administration in healthy male subjects at steady state.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the informed consent form (ICF) and giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Healthy male subjects aged 18 to 45 years inclusive, at the time of signing the ICF, able to tolerate venipuncture.
3. Verified diagnosis of being "healthy" according to results of standard clinical, laboratory and instrumental methods of examination.
4. Body weight ≥50 kg and ≤ 120 kg, Body Mass Index between ≥18.5 and ≤30.0 kg/m2.
5. Non-smokers (for at least 3 months).
6. Subjects should be willing to remain abstinent (refrain from heterosexual intercourse) or use double barrier contraception during participation in the study and for 30 days thereafter. Double-barrier contraceptive method: condom used together with spermicidal foam/gel/film/cream/suppository.

Exclusion Criteria:

1. History or presence of allergies.
2. Known hypersensitivity or intolerance to tamsulosin and/or other alpha1 adreno-receptor antagonists and/or any excipient of the study drugs.
3. History of drug-induced angioedema.
4. History, presence or necessity of glaucoma or cataract surgery.
5. History or presence of acute or chronic diseases of cardiovascular (including arterial hypotension), bronchopulmonary, nervous, endocrine, reproductive systems (including ejaculation disorders), and also diseases of the gastrointestinal tract, liver (including hepatic insufficiency), urinary tract and kidneys (including renal insufficiency), blood, mental diseases; history of convulsive attacks.
6. Acute infectious diseases (e.g. influenza, acute respiratory viral infections incl. COVID-19) less than 4 weeks before the first IMP administration.
7. The presence of any other condition which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results, or the subject's ability to participate in the study.
8. Surgery on the gastrointestinal tract (except appendectomy).
9. Deviations from the normal parameters in clinical blood count analysis, biochemical blood analysis, urinalysis.
10. History or presence of orthostatic hypotension or syncope.
11. Systolic blood pressure measured in a sitting position, less than 100 mmHg or above 130 mmHg and/or diastolic blood pressure below 60 mmHg or above 89 mmHg.
12. Heart rate less than 60 or more than 80 beats per minute.
13. Deviation on the ECG intervals and heart rate or ECG morphology.
14. Positive test results for HIV or hepatitis B or C or syphilis at screening.
15. Positive test result for cotinine in the urine at screening or before randomisation.
16. Positive screen for drugs or alcohol at screening or before randomisation.
17. Known or suspected drug or alcohol abuse as judged by the Investigator.
18. Alcohol consumption more than 10 units of alcohol a week (1 unit equivalent to 200 ml of dry wine or 50 ml of strong alcoholic drinks or 500 ml of beer) during the six months prior to the first administration of the IMP.
19. Intake of xanthine containing substances (e.g., coffee, tea, chocolate, energy drinks, cola) as well as citrus fruits (grapefruit, grapefruit juice etc.) and cranberry (including juices, fruit drinks, etc.) within the last 72 hours before the IMP administration.
20. Administration of medicines that have a significant effect on circulatory dynamics, liver function, etc. (barbiturates, omeprazol, cimetidin, NSAIDs, ACE inhibitors, angiotensin II receptor antagonists, diuretics, etc.) less than 2 months or 5 half-lives (whatever is longer) before screening.
21. The use of depot-forms of any drugs for 3 months or 5 half-lives (whatever is longer) before screening.
22. Use of any prescribed or non-prescribed medication, herbal remedies, vitamins and minerals during the two weeks prior to the first administration of the IMP or longer (at least 5 elimination half-lives) if the medication has a long half-life.
23. Mental, physical and other reasons that do not allow the subjects according to investigator's opinion to assess their behavior adequately, to follow correctly the requirements of the clinical study protocol and to assess the expected risks and possible discomfort.
24. Dehydration (e.g. due to diarrhea, vomiting, or other causes) within the last 48 hours before the IMP administration.
25. Subjects who have been on a special diet (for whatever reason, e.g. vegetarians or hypocaloric diet [less than 1000 cal/day]) during the 28 days prior to the first IMP administration and intention to maintain the diet during the study.
26. Intention to perform excessive physical activities during the trial.
27. Plasma donation within one month of screening or blood donation/blood loss >500 ml within 3 months before screening.
28. Unwillingness or inability to follow the procedures and restrictions outlined in the protocol and the ICF.
29. Participation in another clinical study within 3 months before the first IMP administration.
30. Difficulty swallowing tablets or fasting or consuming standard meals.
31. Any reason in the opinion of the Investigator, would prevent the subject from participating in the study.
32. Scheduled to have vaccination during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Tamsulosin is indicated for the treatment of benign prostatic hyperplasia (BPH). Therefore, only male subjects were included
Enrollment: 33 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss | 7 days
  Maximum plasma concentration at steady state
AUC(0-tau),ss | 7 days
  Area under the curve at steady state
Ctau,ss | 7 days
  Plasma concentration at the end of the dosing interval at steady state

SECONDARY OUTCOMES:
Cavg,ss | 7 days
  Average concentration at steady state
Tmax,ss | 7 days
  Time to maximum plasma concentration at steady state
Cmin,ss | 7 days
  Minimum plasma concentration at steady state
Kel | 7 days
  Terminal rate constant
PTF | 7 Days
  Peak-trough fluctuation over one dosing interval at steady state
T 1/2 | 7 days
  Plasma half life
Swing | 7 days
  (Cmax,ss-Cmin,ss)/ Cmin,ss

OTHER OUTCOMES:
Analysis of adverse events (AE) | 31 days
  Number (%) of subjects with any AE
Analysis of adverse events (AE) | 31 days
  Number (%) of subjects with treatment-related AEs
Analysis of adverse events (AE) | 31 days
  Number (%) of subjects with any serious adverse events (SAE)
Analysis of adverse events (AE) | 31 days
  Number (%) of subjects with treatment-related SAEs
Analysis of adverse events (AE) | 31 days
  Number (%) of subjects discontinued from the study due to AEs

CONTACTS AND LOCATIONS:
Locations (1):
- "Tonus-Les" LLC, Yerevan, Akunk Region, Armenia

IPD SHARING:
Plan to Share IPD: No
No publication in an ICMJE journal is planned

REFERENCES:
- See also: Related Info — https://www.menarini.com/en-us/innovation-research/clinical-trials/clinical-trials-database.html